CLINICAL TRIAL: NCT00582543
Title: MRI/MRSI in Risk Assessment of Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-113
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Physicians; Prostatectomy; Radiotherapy; Therapeutics

ARMS (1):
- eMRI/MRSI (Experimental): Patients will undergo eMRI/MRSI examination. Upon arrival at the MRI suite, patients will be asked to complete a standard MRI screening form. Patients will be scanned in the supine position.
  Interventions: Other: eMRI/MRSI

INTERVENTIONS:
Other: eMRI/MRSI — Patients will undergo eMRI/MRSI examination. All subjects will be asked to administer a Fleet enema on the day of the study in order to reduce the potential for fecal residue to interfere with imaging acquisition and quality. Upon arrival at the MRI suite, patients will be asked to complete a standard MRI screening form. Patients will be scanned in the supine position. The entire eMRI/MRSI study will be performed within 55-60 minutes.
  Other Names: All patients enrolled in the protocol will have clinically indolent disease as; defined by NCCN guidelines. Treatment selection between definitive treatment; and deferred therapy will be decided jointly by the patient and the treating; physician (non-randomized selection). Patients will be treated with radical; prostatectomy (RP) or radiation therapy (RT) or will be placed on deferred; therapy.

SUMMARY:
The purpose of this study is to see if magnetic resonance imaging (MRI) and magnetic resonance spectroscopic imaging (MRSI) can tell which patients with prostate cancer are at a low risk for their cancer growing and spreading. Magnetic resonance methods use magnets and radio waves to take pictures of body structure (MRI) and to measure amounts of important chemicals within the body (MRSI). This study will look at the structural and chemical properties of prostates before undergoing treatment. Hopefully, doctors will be able to use this method before making treatment decisions for patients with newly diagnosed cancer of the prostate. This study will continue our work to assess the value of MRI/MRSI in addressing what is currently one of the greatest clinical challenges in the management of prostate cancer: the identification of low-risk organ-confined prostate cancer that can be managed expectantly with deferred treatment.

DETAILED DESCRIPTION:
In this study, patients with low-risk, organ-confined prostate cancer identified in clinic or prior to their already scheduled standard of care MRI in the Department of Radiology will be approached for the study. Eligible patients will undergo a baseline eMRI/MRSI exam between 6 and 24 weeks following biopsy. Patients will undergo definitive treatment (radical prostatectomy (RP) or radiation therapy (RT)) or will be placed on deferred therapy. Predictor variables will be recorded for each patient after enrollment, before treatment and during treatment follow-up. Patient outcome-disease progression will be determined by long term clinical follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Gleason ≤6 (grade 3 + 3 or lower) biopsy proven prostate cancer
2. Clinically low-risk localized disease as defined by NCCN guidelines (clinical stage T1-T2a, maximum Gleason score 2-6, peak serum PSA level < 10 ng/ml)
3. No evidence of disseminated disease (bone or lymph node metastases)
4. Treatment-radical prostatectomy, radiation therapy, or deferred therapy-will be at MSKCC
5. Willingness to undergo serial surveillance TRUS-guided prostate biopsies and eMRI/MRSI examination at MSKCC if placed on deferred therapy protocol
6. In the surgical cohort, RP (radical prostatectomy) is scheduled to occur within six months of eMRI/MRSI study

Exclusion Criteria:

1. Prior treatment (e.g. with hormonal therapy, radical prostatectomy, radiation therapy or cryosurgery)
2. Inability to give informed consent because of age, general medical or psychiatric condition, or physiologic status
3. Presence of known contraindication to eMRI
4. Unwillingness or inability to undergo placement of endorectal MR coil or ultrasound probe. As is the case for a standard MR exam, the presence of a pacemaker or aneurysm clips could pose a risk to patients, making them unable to have an eMRI, and therefore unable to participate in this study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2005-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
In a population of patients designated as clinically indolent by NCCN guidelines, we will evaluate the ability of eMRI/MRSI to predict pathologically indolent cancer. eMRI/MRSI findings will be compared with step-section pathology. | October 2010

SECONDARY OUTCOMES:
In the patients who are identified as harboring indolent prostate cancer by both clinical guidelines and eMRI/MRSI, clinical progression of disease will be evaluated in a cohort of patients receiving deferred therapy. | October 2010
We will explore whether eMRI/MRSI markers of progression correlate with clinical markers of progression. | October 2010
  Patients undergoing deferred treatment will undergo followup eMRI/MRSI exams before surveillance biopsies, beginning approximately 12-18 months after confirmatory biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Hedvig Hricak, M.D., Ph.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org